CLINICAL TRIAL: NCT02496026
Title: Transcranial Direct Current Stimulation and Robotic Therapy in Upper Limb Motor Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auxilium Vitae Volterra (Other)
Responsible Party: Principal Investigator, federico posteraro, Medical Doctor, Auxilium Vitae Volterra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RN20141
Record Dates: First submitted 2015-07-02; First posted 2015-07-14 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2019-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS plus wrist robot therapy (Experimental): In addition to standard rehabilitation treatment Group A will perform daily sessions of wrist robot-assisted treatment in combination with tDCS (30 minutes). During first 20 min of each session the patient receives a direct current stimulation through surface sponge electrodes (35 cm2), 2 milliampere intensity: the anodal electrode is placed on presumed lesional area, the cathodal electrode is placed on the controlateral orbital bone.
  Interventions: Device: tDCS plus wrist robot therapy
- Sham tDCS plus wrist robot therapy (Sham Comparator): Group B is treated as Group A, but tDCS, even if the cap is applied on the patient head, is not activated and no current is delivered.
  Interventions: Device: Sham tDCS plus wrist robot therapy

INTERVENTIONS:
Device: tDCS plus wrist robot therapy — Patients receive robotic rehabilitation session while tDCS stimulator is switched on
  Arms: tDCS plus wrist robot therapy
Device: Sham tDCS plus wrist robot therapy — Patients receive robotic rehabilitation session while tDCS stimulator is switched off.
  Arms: Sham tDCS plus wrist robot therapy

SUMMARY:
The objective of the study is to evaluate the effectiveness of transcranial direct current stimulation (tDCS) integrated with wrist robot-assisted treatment. In detail, the anodal stimulation on the impaired hemisphere will be used associated with a robotic treatment.

DETAILED DESCRIPTION:
As for transcranial direct current stimulation a HDC kit (ATES/EB NEURO, Firenze, Italy) will be used as device. It is a new device generation of stimulator able to provide an effective stimulation pattern.

As robotic device the InMotion wrist robot (Interactive Motion Technologies Inc., Watertown, MA, USA) will be used. It is an end-effector robotic device able to assist as needed the wrist movements.

ELIGIBILITY:
Inclusion Criteria:

1. persons affected by first supratentorial stroke, whose onset time is 25±7 days;
2. upper limb hemiparesis;
3. cognitive and speech abilities sufficient to understand instructions and to provide informed consent;
4. absence of intense pain due to passive wrist mobilization assessed by VAS < 3 (range 0-10);
5. ability to provide written informed consent.

Exclusion Criteria:

1. previous epilepsy seizures;
2. severe electroencephalographic anomalies;
3. previous neurosurgery interventions involving metallic elements placement;
4. ongoing anticonvulsant drugs treatment
5. inability to keep sitting posture;
6. severe sensory deficits;
7. general clinical complication preventing delivery of rehabilitation treatment.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the motor impairment as assessed by the Fugl-Meyer Motor Assessment Scale (upper extremity subsection) | 6 weeks
  Impairment level measure according to ICF

SECONDARY OUTCOMES:
Change from Baseline in the motor impairment as assessed by the Fugl-Meyer Motor Assessment Scale (upper extremity subsection) | 6 months
  Impairment level measure according to ICF
Change from Baseline in the upper limb functional and motor abilities as assessed by the Motricity Index | 6 weeks
  Impairment level measure according to ICF
Change from Baseline in the upper limb functional and motor abilities as assessed by the Motricity Index | 6 months
  Impairment level measure according to ICF
Change from Baseline in the upper limb spasticity as assessed by the Modified Ashworth Scale | 6 weeks
  Impairment level measure according to ICF
Change from Baseline in the upper limb spasticity as assessed by the Modified Ashworth Scale | 6 months
  Impairment level measure according to ICF
Change from Baseline in the unilateral gross manual dexterity as assessed by the Block and Box test | 6 weeks
  Activities level measure according to ICF
Change from Baseline in the unilateral gross manual dexterity as assessed by the Block and Box test | 6 months
  Activities level measure according to ICF

CONTACTS AND LOCATIONS:
Overall Officials: Federico Posteraro, MD, Principal Investigator — Auxilium Vitae Rehabilitation Centre; Stefano Mazzoleni, PhD, Study Director — The BioRobotics Institute, Scuola Superiore Sant'Anna
Locations (1):
- Auxilium Vitae Rehabilitation Centre, Volterra, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehrholz J, Platz T, Kugler J, Pohl M. Electromechanical and robot-assisted arm training for improving arm function and activities of daily living after stroke. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006876. doi: 10.1002/14651858.CD006876.pub2. PMID 18843735
- [Background] Floel A, Rosser N, Michka O, Knecht S, Breitenstein C. Noninvasive brain stimulation improves language learning. J Cogn Neurosci. 2008 Aug;20(8):1415-22. doi: 10.1162/jocn.2008.20098. PMID 18303984
- [Background] Kang EK, Baek MJ, Kim S, Paik NJ. Non-invasive cortical stimulation improves post-stroke attention decline. Restor Neurol Neurosci. 2009;27(6):645-50. doi: 10.3233/RNN-2009-0514. PMID 20042788
- [Background] Marangolo P, Marinelli CV, Bonifazi S, Fiori V, Ceravolo MG, Provinciali L, Tomaiuolo F. Electrical stimulation over the left inferior frontal gyrus (IFG) determines long-term effects in the recovery of speech apraxia in three chronic aphasics. Behav Brain Res. 2011 Dec 1;225(2):498-504. doi: 10.1016/j.bbr.2011.08.008. Epub 2011 Aug 12. PMID 21856336
- [Background] Fiori V, Coccia M, Marinelli CV, Vecchi V, Bonifazi S, Ceravolo MG, Provinciali L, Tomaiuolo F, Marangolo P. Transcranial direct current stimulation improves word retrieval in healthy and nonfluent aphasic subjects. J Cogn Neurosci. 2011 Sep;23(9):2309-23. doi: 10.1162/jocn.2010.21579. Epub 2010 Oct 14. PMID 20946060
- [Background] Hesse S, Waldner A, Mehrholz J, Tomelleri C, Pohl M, Werner C. Combined transcranial direct current stimulation and robot-assisted arm training in subacute stroke patients: an exploratory, randomized multicenter trial. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):838-46. doi: 10.1177/1545968311413906. Epub 2011 Aug 8. PMID 21825004
- [Derived] Mazzoleni S, Tran VD, Dario P, Posteraro F. Effects of Transcranial Direct Current Stimulation (tDCS) Combined With Wrist Robot-Assisted Rehabilitation on Motor Recovery in Subacute Stroke Patients: A Randomized Controlled Trial. IEEE Trans Neural Syst Rehabil Eng. 2019 Jul;27(7):1458-1466. doi: 10.1109/TNSRE.2019.2920576. Epub 2019 Jun 3. PMID 31170077